CLINICAL TRIAL: NCT02042612
Title: Pharmacokinetic Study of 48-hour Sevoflurane Inhalation Using a Disposable Delivery System (AnaConDa©) in Obese ICU Patients
Acronym: CISEVOB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0176; 2010-020044-35
Record Dates: First submitted 2014-01-14; First posted 2014-01-23 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Obesity
Keywords: Pharmacokinetics; Sevoflurane; Obesity; Sedation; ICU patients
MeSH Terms: conditions — Obesity | interventions — Intensive Care Units

ARMS (1):
- sevoflurane (Experimental): Determination of plasmatic concentrations of sevoflurane at different times of a 48h sedation of sevoflurane in obese ICU patients
  Interventions: Drug: Sedation with sevoflurane during 48-hr in ICU

INTERVENTIONS:
Drug: Sedation with sevoflurane during 48-hr in ICU
  Other Names: Determination of plasmatic concentrations of sevoflurane at different times of a 48h sedation of sevoflurane in obese ICU patients

SUMMARY:
Describing a pharmacokinetic model of 48-h sevoflurane sedation in obese ICU patients

DETAILED DESCRIPTION:
Prospective clinical monocentric study in ICU with sedated ventilated obese patients with sevoflurane during 48 h with the AnaConda® system, establishing pharmacokinetic model of sévoflurane and its metabolites (hydroxyfluroisopropanol, fluoride)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ventilated more than 48 h Stable respiratory and hemodynamic conditions Consent of patients or family Arterial line BMI >30

Exclusion Criteria:

* Acute kidney injury BMI <30 Sevoflurane anaphylaxia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Determination of plasmatic concentrations of sevoflurane before using AnaConda® system | at 5min, 60 min, 24 hrs and just before the end of sedation.

SECONDARY OUTCOMES:
Determination of plasmatic concentrations of HFIP and fluoride before using AnaConda® system | at 5min, 60 min, 24 hrs and just before the end of sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France